CLINICAL TRIAL: NCT00797238
Title: DNA Repair Genes and Outcomes in Patients With Stage III NSCLC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Chao-Chi Ho, National Taiwan University Hospital
Other Study IDs: 200709017R
Record Dates: First submitted 2008-07-09; First posted 2008-11-25 (Estimated); Last update posted 2010-07-15 (Estimated); Status verified 2010-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Chemotherapy
Keywords: Gene Expression; Carcinoma, Non-Small-Cell Lung; Chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — lung cancer tissue before and after treatment
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- NSCLC stage III: Taiwanese NSCLC patients with stage III

INTERVENTIONS:
Other:  — No intervention in this study
  Other Names: No intervention in this study

SUMMARY:
The studied materials contains surgically specimens of two groups of patiens with non-small cell lung cancer who have received two regimens of induction (neoadjuvant) chemotherapy before tumor resection. Pathological specimens of pre-chemotherapy and post-chemotherapy whatever retrievable will be collected. The protein ad RNA expression of DNA repair genes (ERCC1, ERCC2, XRCC1, XRCC3, BRCA1 and RRM1) as well as DNA polymorphisms of these genes will be studied, and will be correlate with the treatment response and outcome of the patients. The aims of this study include:

1. To identify the expression status of the above DNA repair genes in Taiwanese NSCLC patients.
2. To correlate the expression, as well as DNA polymorphism of each DNA repair gene in treatment response to two differenct chemotherapeutic regimens.
3. To correlate the expression, as well as DNA polymorphism of each DNA repair gene in the outcome of stage III NSCLC patients.
4. To explore whether platinum based chemotherapy will change the expression status of DNA repair gene and if indeed changed, whether this would influence the outcome of the patients

DETAILED DESCRIPTION:
Patients with clinical stage IIIA N2 non-small cell lung cancer (NSCLC) have a 5-year survival rate of 10% to 15%, much worse than those of earlier stages of disease. The use of pre-operative (neo-adjuvant) chemotherapy has been shown to be beneficial in several studies.1 However, the precise chemotherapeutic regimen for neoadjuvant therapy remains an open question.

The treatment response and toxicity of chemotherapy vary widely among and within individuals, and races. Recently, molecular predictive markers may help to identify who may benefit from individual therapy. Many evidence shows that the level of ERCC1 (an excision nuclease within the nucleotide excision repair pathway) is important for the repair of platinum-DNA adducts and the response to platinum-based chemotherapy.2-5 Not only by measuring protein and mRNA expression, studies addressed on the polymorphism of ERCC1(118 C/T and C8092A) had demonstrated impact on survival of chemotherapy-treated NSCLC patients6,7. XPD/ERCC2 (xeroderma pigmentosum group D/excision repair cross-complementing group 2) 8, XRCC1 (X-ray repair cross-complementing group 1) and XRCC3 (X-ray repair cross-complementing group 3) are another three proteins involving NER, serving as prognostic factor of survival.9 BRCA1 is a protein participating in recombinant repair (RR) and is stronge predictive marker of chemotherapy response. BRCA1 functions as a differential modulator of survival with cisplatin and antimicrotubule drugs (paclitaxel, docetaxel and vinorelbine). Low level of BRCA1 enhance cisplatin activity but lead to resistance to paclitaxel, docetaxel and vinorelbine, whereas the opposite phenomenon is observed in the presence of normal or high levels of BRCA1. In contract, BRCA1 levels do not influence the effect of gemcitabine10. On the contrary, RRM1 (ribonucleotid reductase subunit M1) is involved in gemcitabine metabolism and DNA repair after chemotherapy damage, and increased RRM1 mRNA expression has been related to gemcitabine resistance in NSCLC11. All these DNA repair genes participate the pathogenesis, mechanism of chemotherapeutic resistance and outcome of lung cancer patients.

Previously, a joint study done by NTUH and VGH Taipei used gemcitabine and cisplatin as induction chemotherapy to treat 52 patient with stage III NSCLC, 36 were operable and 18 were completely resected.12 From 2004 till now, a prospective study has been performed in NTUH using docetaxel and cisplatin as neoadjuvant regimen to treat patients with stage IIIA (N2) non-small cell lung cancer. Up to now, more than 40 patients were enrolled, all of them have received tumor sampling before chemotherapy and more 90% received operation with their tumor resected. The tissue specimens are valuable as all these patients had received protocolized treatment, with filed detailed clinical information collected systematically. All the peroperative biopsied and operatively resected tumor tissues are available in paffin-embedded block, some in frozen tissue stock, we plan to study the DNA polymorphism, protein and RNA expression of the above-mentioned DNA repair genes in these two series of patients.

ELIGIBILITY:
Inclusion Criteria:

* NSCLC patients with stage III in NTUH
* Recieved neoadjuvant chemotherapy and received operation

Exclusion Criteria:

* Patients who did not received chemotherapy or they did not receive operation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Taiwanese NSCLC patients with stage III
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-09; Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Change of the expression status of the DNA repair genes after chemotherapy in Taiwanese NSCLC patients | before and after chemotherapy

SECONDARY OUTCOMES:
Relationship between change of the expression status of the DNA repair genes after chemotherapy and clinical outcome

CONTACTS AND LOCATIONS:
Overall Officials: Chao-Chi Ho, Ph.D., Principal Investigator — Department of Internal Medicine and Emergency Medicine, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan